CLINICAL TRIAL: NCT03106025
Title: Use of Ocular Point of Care Ultrasound in Diagnosing Retinal Detachment in the Emergency Department: A Prospective Study.
Brief Title: Use of Ocular Point of Care Ultrasound in Diagnosing Retinal Detachment in the Emergency Department
Acronym: RDOcularUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Tze Lyn Stephanie Tseeng, Emergency Medicine Specialist, Loma Linda University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 5170078
Record Dates: First submitted 2017-04-04; First posted 2017-04-10 (Actual); Results first posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-09

CONDITIONS: Retinal Detachment
MeSH Terms: conditions — Retinal Detachment | interventions — Ultrasonography

STUDY DESIGN:
Masking Description: ophthalmologists will be blinded to the ultrasound result and formal ophthalmology assessment will be compared to the ultrasound assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Patients Receiving Ophthalmology Assessment (Active Comparator): Number of subjects with retinal detachment per formal ophthalmology assessment. This assessment is a composite measurement which includes the following chief complain, primary impression, right visual acuity, left visual, acuity, ultrasound diagnosis, diagnosis changed, ophthalmology diagnosis.
  Interventions: Device: Ultrasound; Other: Ophthalmology Assessment
- Ocular Ultrasound (Experimental): Each participant will receive an ocular ultrasound which poses minimal to no harm to the participant and the ultrasound results compared to final diagnosis
  Interventions: Device: Ultrasound; Other: Ophthalmology Assessment

INTERVENTIONS:
Device: Ultrasound — Each participant will receive an ocular ultrasound which poses minimal to no harm to the participant and the ultrasound results compared to final diagnosis.
Other: Ophthalmology Assessment — Number of subjects with retinal detachment per formal ophthalmology assessment. This assessment is a composite measurement which includes the following chief complain, primary impression, right visual acuity, left visual, acuity, ultrasound diagnosis, diagnosis changed, ophthalmology diagnosis.

SUMMARY:
The study is collecting data along with other academic institutions regarding the accuracy of ocular ultrasound in diagnosing retinal detachment.

DETAILED DESCRIPTION:
This is a prospective, cross-sectional study to assess the utility of point of care ultrasound in the diagnosis of ocular complaints in the emergency department (ED) with specific focus on the accuracy of diagnosis when compared to that of a blinded ophthalmologist. Ocular complaints represent between 2% and 3% of ED visits (Walker et al, 2011). This percentage may include vision-threatening diagnoses including retinal detachment, which can occur in 3-4% of patients presenting with ocular complaints (Alotaibi et al, 2011). However, the equipment and expertise required to adequately assess for conditions such as retinal detachment are limited in busy emergency departments due to the time consuming and challenging nature of the examination. Incorporating the use of an ultrasound could provide a more available, focused, and timely assessment.

ELIGIBILITY:
Inclusion Criteria:

Clinical suspicion for retinal detachment Age >18 years of age Ophthalmology Consult

Exclusion Criteria:

Concurrent ocular trauma Ruptured globe Pregnancy < 18 years of age No ophthalmology consult

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2018-03-25 (Actual); Study Completion 2018-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tze Lyn S Tseeng, MD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University Health, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: Yes
shared across other sites that are pooling data across redcap.
Supporting Information: CSR
Time Frame: February 5, 2018 through March 25, 2018 (approximately 8 weeks)
Access Criteria: Participant sites maintaining a study redcap account

REFERENCES:
- [Background] Walker RA, Adhikari S. Chapter 236 p1517-1549. Eye Emergencies. In: Tintinali JE, Kelen GD, Stapczynski JS, eds. Tintinalli's Emergency Medicine: A Comprehensive Study Guide. 7th ed. New York: McGraw-Hill; 2011.
- [Background] Alotaibi AG, Osman EA, Allam KH, Abdel-Rahim AM, Abu-Amero KK. One month outcome of ocular related emergencies in a tertiary hospital in Central Saudi Arabia. Saudi Med J. 2011 Dec;32(12):1256-60. PMID 22159380
- [Background] Lizzi FL, Coleman DJ. History of ophthalmic ultrasound. J Ultrasound Med. 2004 Oct;23(10):1255-66. doi: 10.7863/jum.2004.23.10.1255. No abstract available. PMID 15448314
- [Background] Coleman DJ, Konig WF, Katz L. A hand-operated, ultrasound scan system for ophthalmic evaluation. Am J Ophthalmol. 1969 Aug;68(2):256-63. doi: 10.1016/0002-9394(69)94068-9. No abstract available. PMID 4307960
- [Background] Vrablik ME, Snead GR, Minnigan HJ, Kirschner JM, Emmett TW, Seupaul RA. The diagnostic accuracy of bedside ocular ultrasonography for the diagnosis of retinal detachment: a systematic review and meta-analysis. Ann Emerg Med. 2015 Feb;65(2):199-203.e1. doi: 10.1016/j.annemergmed.2014.02.020. Epub 2014 Mar 27. PMID 24680547
- [Background] Blaivas M, Theodoro D, Sierzenski PR. A study of bedside ocular ultrasonography in the emergency department. Acad Emerg Med. 2002 Aug;9(8):791-9. doi: 10.1111/j.1553-2712.2002.tb02166.x. PMID 12153883
- [Background] Shinar Z, Chan L, Orlinsky M. Use of ocular ultrasound for the evaluation of retinal detachment. J Emerg Med. 2011 Jan;40(1):53-7. doi: 10.1016/j.jemermed.2009.06.001. Epub 2009 Jul 21. PMID 19625159
- [Background] Yoonessi R, Hussain A, Jang TB. Bedside ocular ultrasound for the detection of retinal detachment in the emergency department. Acad Emerg Med. 2010 Sep;17(9):913-7. doi: 10.1111/j.1553-2712.2010.00809.x. PMID 20836770
- [Background] Teismann N, Lenaghan P, Nolan R, Stein J, Green A. Point-of-care ocular ultrasound to detect optic disc swelling. Acad Emerg Med. 2013 Sep;20(9):920-5. doi: 10.1111/acem.12206. PMID 24050798
- [Background] Blaivas M, Theodoro D, Sierzenski PR. Elevated intracranial pressure detected by bedside emergency ultrasonography of the optic nerve sheath. Acad Emerg Med. 2003 Apr;10(4):376-81. doi: 10.1111/j.1553-2712.2003.tb01352.x. PMID 12670853
- [Background] Tayal VS, Neulander M, Norton HJ, Foster T, Saunders T, Blaivas M. Emergency department sonographic measurement of optic nerve sheath diameter to detect findings of increased intracranial pressure in adult head injury patients. Ann Emerg Med. 2007 Apr;49(4):508-14. doi: 10.1016/j.annemergmed.2006.06.040. Epub 2006 Sep 25. PMID 16997419
- [Background] Geeraerts T, Merceron S, Benhamou D, Vigue B, Duranteau J. Non-invasive assessment of intracranial pressure using ocular sonography in neurocritical care patients. Intensive Care Med. 2008 Nov;34(11):2062-7. doi: 10.1007/s00134-008-1149-x. Epub 2008 May 29. PMID 18509619
- [Background] Kimberly HH, Shah S, Marill K, Noble V. Correlation of optic nerve sheath diameter with direct measurement of intracranial pressure. Acad Emerg Med. 2008 Feb;15(2):201-4. doi: 10.1111/j.1553-2712.2007.00031.x. PMID 18275454
- [Background] Kang TL, Seif D, Chilstrom M, Mailhot T. Ocular ultrasound identifies early orbital cellulitis. West J Emerg Med. 2014 Jul;15(4):394. doi: 10.5811/westjem.2014.4.22007. No abstract available. PMID 25035741

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Receiving Ultrasound: Enrolled participants will receive a bedside ocular ultrasound of the affected eye and the ultrasound will be compared with the ophthalmologist diagnosis. The participant's medical record will also be reviewed for information regarding demographics, complications, and outcomes.
  Ultrasound: Each participant will receive an ocular ultrasound which poses minimal to no harm to the participant and the ultrasound results compared to final diagnosis.
Period: Overall Study
Arm/Group | Patients Receiving Ultrasound
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Same criteria as participant flow assignment.
Arm/Group | Patients Receiving Ultrasound
Number analyzed (Participants) | 5
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 52 [52 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Retinal detachment diagnosis [Number; unit: participants] — Subjects diagnosed with retinal detachment or vitreous detachment.
  participants | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Retinal Detachment Per Ultrasound Assessment
Description: Number of Participants with retinal detachment per ocular ultrasound results
Time Frame: at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Receiving Ultrasound
Number analyzed (Participants) | 5
Participants | 5

ADVERSE EVENTS:
Time Frame: at baseline
Description: These subjects are seen on a one time bases in the emergency department and so adverse events, if they are occur, are collected at baseline.
Arm/Group | Patients Receiving Ultrasound
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

LIMITATIONS AND CAVEATS:
The info entered reflects one Emergency Department site.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-08-21): https://cdn.clinicaltrials.gov/large-docs/25/NCT03106025/Prot_SAP_002.pdf
  • Informed Consent Form (2017-08-21): https://cdn.clinicaltrials.gov/large-docs/25/NCT03106025/ICF_003.pdf